CLINICAL TRIAL: NCT01024907
Title: Proton Radiation for Low Grade Gliomas
Brief Title: Proton Beam Radiation Therapy in Treating Patients With Low Grade Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 08309; NCI-2009-01442
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Adult Brain Tumor; Adult Brain Stem Glioma; Adult Diffuse Astrocytoma; Adult Ependymoma; Adult Grade II Meningioma; Adult Melanocytic Lesion; Adult Meningeal Hemangiopericytoma; Adult Mixed Glioma; Adult Oligodendroglioma; Adult Pineal Gland Astrocytoma; Adult Pineocytoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Ependymoma; Glioma; Oligodendroglioma; Pinealoma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo proton beam radiation therapy for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: proton beam radiation therapy; Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Radiation: proton beam radiation therapy — Undergo radiation
Procedure: quality-of-life assessment — Ancillary study
Other: questionnaire administration — Ancillary study

SUMMARY:
RATIONALE: Specialized radiation therapy, such as proton beam radiation therapy, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase I/II trial is studying the best way to give proton beam radiation therapy and to see how well it works in treating patients with low grade gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of proton beam radiation therapy in patients with low grade gliomas. (Phase I)

SECONDARY OBJECTIVES:

I. To assess late complications from irradiation using proton beam therapy in place of conventional photon beam therapy for the treatment of low grade gliomas. (Phase II) II. To assess acute side effects from irradiation using proton beam therapy in place of conventional photon beam therapy for the treatment of low grade gliomas. (Phase II) III. To compare the dose distribution to tumor and surrounding normal structures using DVH's (Dose Volume Histograms) generated from the proton plan used to treat the patient and the photon plan generated for comparison purposes. (Phase II) IV. To monitor the rates of local control, overall and disease specific survival using proton radiotherapy. (Phase II) V. To evaluate the time to progression of low grade gliomas treated with protons. (Phase II) VI. To evaluate the incidence and severity of fatigue in low grade glioma treated with protons. (Phase II) VII. To evaluate the effect of proton beam radiation on neurocognitive outcome in patients with low grade glioma. (Phase II) VIII. To evaluate the quality of life in patients treated for low grade glioma. (Phase II)

OUTLINE: Patients undergo proton beam radiation therapy for 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion

* Patients with histologically confirmed diagnosis of low grade glioma of the CNS
* Patients with WHO grade II; may be symptomatic; including patients who are being followed and have radiographic expression
* Patients must have a Karnofsky Performance Status of >= 60
* Patients must be able to provide informed consent
* Patients must have adequate bone marrow function:

  1. WBC >= 4000/mm^3
  2. platelets >= 100,000 mm^3
* Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms or other barrier methods etc); Hysterectomy or menopause must be clinically documented

Exclusion

* Patients who have had prior or simultaneous malignancies within the past two years (other than cutaneous squamous or basal cell carcinoma, melanoma in situ or thyroid carcinoma)
* Patients with the following histologies:

gliomatosis cerebrei, WHO III or IV gliomas

* Patients who have had any prior Radiation treatment
* Patients who have had any chemotherapy administered within 30 days of the planned radiation treatment start date
* Pregnant women, women planning to become pregnant and women that are nursing
* Patients who are actively being treated on any other therapeutic research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-12-17 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Feasibility (phase I)
Acute toxicity as assessed by NCI CTC version 3.0 (phases I and II) | 60 days (phase I) or 90 days (phase II) from completion of radiation therapy

SECONDARY OUTCOMES:
Late toxicity as graded according to the RTOG/EORTC late morbidity scoring system (phases I and II)
Fatigue as assessed by the Brief Fatigue Inventory (phases I and II) | Pre-radiation, mid-treatment, and post-radiation; at 3, 6, 9, and 12 months post-radiation; and then every 6 months
Cumulative total dose to normal brain tissue (phase II)
Progression-free survival (phases I and II)
Overall survival (phases I and II)
Adverse events as assessed by NCI CTCAE version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lustig, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Maquilan G, Grover S, Alonso-Basanta M, Lustig RA. Acute toxicity profile of patients with low-grade gliomas and meningiomas receiving proton therapy. Am J Clin Oncol. 2014 Oct;37(5):438-43. doi: 10.1097/COC.0b013e31827de86b. PMID 23388559